CLINICAL TRIAL: NCT01899196
Title: EPICARDIAL ADIPOSE TISSUE AND CORONARY RISK IN HIV-INFECTED PATIENTS
Acronym: ANRS EP 52
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ANRS EP 52 PIECVIH
Record Dates: First submitted 2013-07-02; First posted 2013-07-15 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Hiv Infection
Keywords: Cardiac surgery
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- no Arm (Other)
  Interventions: Biological: blood sampling,

INTERVENTIONS:
Biological: blood sampling,

SUMMARY:
Protocol date and version RCB Id : 2013-A00547-38

Etude ANRS EP 52 PIECVIH Title of Study: EPICARDIAL ADIPOSE TISSUE AND CORONARY RISK IN HIV-INFECTED PATIENTS

Short title - PIECVIH study

Sponsor French National Institute for Health and Medical Research - French national agency for research on AIDS and viral hepatitis (Inserm-ANRS)

Coordinating Investigator Pr Franck BOCCARA Service de Cardiologie, Hôpital St Antoine INSERM UMRS 938 Paris, UPMC, Institut hospitalo-Universitaire- Institute of Cardiometabolism and Nutrition (IHU-ICAN) 184, rue du Faubourg Saint-Antoine 75571 PARIS Cedex 12 Tél. : 01 49 28 24 49 - Fax : 01 49 28 26 83 Courriel : franck.boccara@sat.aphp.fr

Participating country: France

Objectives Principal objective To compare the inflammatory profile of the epicardial adipose tissue (EAT) between people living with and without HIVwho present with coronary heart disease and will undergo a coronary artery bypass graft (CABG)

Secondary objectives

* To compare the volume of EAT between people living with and without HIV who present with coronary heart disease
* To evaluate the relationship between the abnormalities of the expression profiles of the adipocytokines and cytokines with the atherosclerotic lesions.
* To evaluate the relationship between the abnormalities of the expression profiles of the adipocytokines and cytokines of the EAT with the circulating levels and metabolic parameters.
* To compare the histological and inflammatory profiles of the EAT with the subcutaneous adipose tissue for each patient individually.

Methodology multicentric, comparative study

Estimated enrollment 31 participants in total

1. st group of- 15 people living with HIV undergoing CABG (coronary heart disease HIV+ group)
2. nd group of- 16 people without HIV- undergoing CABG (coronary heart disease HIV- group) People without HIV-will be matched to people living with HIV+ by : age (± 5 years) and sex Outcomes

Primary outcome:

Comparative analysis of the inflammatory profile of the EAT : expression profile of the pro and anti inflammatory cytokines and adipokines within the EAT in both groups of participants : coronary heart disease HIV+ and HIV- groups

Secondary outcomes :

* Determination of the EAT volume by echocardiography and cardiac scanner for both groups
* Macroscopic profile of the EAT : adipocytes, fibrosis, endothelial cell density)
* RT-PCR analyses : renin, adiponectine, PPARɣ
* Comparatison of the inflammatory and macroscopic profiles between the EAT and the subcutaneous adipose tissue in the two groups by ARN messagers analysis.

Eligibility Inclusion criteria HIV+ group

* Men or women above the age of 18 years old, HIV1 seropositive for more than 6 months
* Individual undergoing, for the first time, cardiac surgery for CABG
* Affiliated with a social security regimen (the AME is not a social security regimen)
* Signed the consent form

HIV- group

* Men or women above the age of 18 years old, HIV seronegative
* Individuals undergoing, for the first time, cardiac surgery for CABG
* Affiliated with a social security regimen (the AME is not a social security regimen)
* Signed the consent form

Non-inclusion criteria History of surgery for CBAG and/or congenital heart defect- being under the tutorship or guardianship of the state or in custody of the justice system.

Statistical methods Categorical variables will be compared using Fisher's exact test. Continuous variables will be compared using the Student's t-test (parametric) and the Wilcoxon-Mann-Whitney test (non-parametric) as appropriate considering the data distribution. (statistical analysis software STATA 11 (StataCorp, Texas, USA))

Provisional study planning and timetable Study start date: July 2013 Enrollment period: 32 months Subject participation duration: 24 hours Total study duration: 32 months Estimated study completion date: end of March 2016

ELIGIBILITY:
Inclusion Criteria:

VIH + GROUP:

* Men or women > 18 years old, HIV1 + for more than 6 months
* Planned first cardiac surgery for CABG

VIH - GROUP:

* Men or women > 18 years old,
* Planned first cardiac surgery for CABG

Exclusion Criteria:

- History of cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
comparison of the inflammatory profile of the epicardial adipose (EAT) tissue between HIV-infected and uninfected patients undergoing cardiac surgery for coronary artery bypass graft (CABG) | day 1

SECONDARY OUTCOMES:
comparison the volume of EAT between HIV-infected and uninfected patients undergoing cardiac surgery | day 1
Evaluation of the relations between the adipocytokines and cytokines profile in the EAT and in the systemic circulation. | day 1
Comparison of the histological and inflammatory profiles of the EAT and the subcutaneous adipose tissue of each patients. | day 1
Evaluation of the relations between the adipocytokines and cytokines profile in the EAT and coronary artery lesions. | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pascal LEPRINCE, Principal Investigator — Hôpital La Pitié Salpétrière Paris
Locations (1):
- Hospital St Antoine, Paris, France